CLINICAL TRIAL: NCT01609855
Title: Does Hyoscine N-butylbromide Administered During Colonoscopy Increase the Polyp Detection Rate? a Randomized, Single Center, Double Blind, Placebo-controlled Study
Brief Title: Does the Hyoscine N-Butylbromide Administered During Colonoscopy Increase the Adenoma Detection Rate?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Emanuele Rondonotti, Principal investigator, Valduce Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: HBB-1
Record Dates: First submitted 2012-05-07; First posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Colonic Adenomas
Keywords: Adenoma Detection Rate; Anti-spasmotic drug
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- HBB- Hioscine Butyl Bromide (Experimental)
  Interventions: Drug: Hyoscine Butyl Bromide 20mg/2 ml i.v.
- Placebo arm (Placebo Comparator)
  Interventions: Drug: Saline 2 ml i.v.

INTERVENTIONS:
Drug: Hyoscine Butyl Bromide 20mg/2 ml i.v. — Hyoscine Butyl Bromide 20mg/2 ml i.v.is administered at time of caecal intubation
  Other Names: Buscopan: Hyoscine Butyl Bromide 20mg/2 ml i.v.
  Arms: HBB- Hioscine Butyl Bromide
Drug: Saline 2 ml i.v. — Administration of Saline 2 ml at time of caecal intubation
  Other Names: Saline
  Arms: Placebo arm

SUMMARY:
The primary aim of the study was to test if the administration of Hyoscine Butyl Bromide, at time of caecal intubation, increases the adenoma detection rate.

DETAILED DESCRIPTION:
Outpatients referred for colonoscopy were screened for possible enrollment. Exclusion criteria included: glaucoma, benign prostatic hyperplasia or urinary obstruction, previous intestinal resection, ongoing therapy with tricyclic antidepressants, chronic renal failure and history of IBD. Eligible patients were randomized to receive either 20 mg/2ml of HBB i.v. or 2ml of saline i.v.; both the endoscopist and the patient were blind to the administered drug. The endoscopist was asked to inspect the right, transverse and left colon for at least 2 min for each segment. The number, size and location of polyps were recorded as well as the occurrence episodes of tachycardia (defined as bpm>140). As indirect estimation of the amount of air retained in the abdomen at the end of the procedure, the DAC (difference in the abdominal circumference measured before and after colonoscopy) was also calculated. At discharge (at least 1 hour after colonoscopy) the bloating perceived by the patient was measured by means of a VA scale (range 0-100).

ELIGIBILITY:
Inclusion Criteria:

* outpatients referred for colonoscopy

Exclusion Criteria:

* glaucoma
* benign prostatic hyperplasia or urinary obstruction
* previous intestinal resection,
* ongoing therapy with tricyclic antidepressants
* chronic renal failure
* history of IBD
* participation other studies
* unsedated colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Effect of Hyoscine Butyl Bromide on Adenoma Detection Rate (ADR) | 5 months

SECONDARY OUTCOMES:
Tolerability of HBB | this outcome will be evaluated at the end of colonoscopy
  As indirect estimation of the amount of air retained in the abdomen at the end of the procedure, the DAC (difference in the abdominal circumference measured before and after colonoscopy) was also calculated. At discharge (at least 1 hour after colonoscopy) the bloating perceived by the patient was measured by means of a VA scale (range 0-100).

CONTACTS AND LOCATIONS:
Overall Officials: Spinzi Giancarlo, MD, Study Director — Gastroenterology Unit, Ospedale Valduce, Como, Italy.; Franco Radaelli, MD, Study Chair — Gastroenterology Unit, Ospedale Valduce, Como. Italy.; Emanuele Rondonotti, MD, Principal Investigator — Gastroenterology Unit, Ospedale Valduvce, Como. Italy.
Locations (1):
- Ospedale Valduce, Como, Italy